CLINICAL TRIAL: NCT02032563
Title: Study of the (Intravenously Injected) Indocyanine Green Distribution in Tumour Bearing Breasts and in Axillary Pieces of Dissection of Patients Who Have Received Neoadjuvant Therapy for Histologically Proven Mammary Cancer
Brief Title: Study of the ICG Distribution in Breast Tumours or in Axillary Lymph Nodes of Patients After Neoadjuvant Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BR-ICG-IV-NACT
Record Dates: First submitted 2014-01-02; First posted 2014-01-10 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
Keywords: neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Indocyanine Green (Experimental): intravenous injection of 0.25mg/kg Indocyanine Green just before surgery
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — intravenous injection of 0.25mg/kg Indocyanine Green just before the surgery
  Other Names: ICG

SUMMARY:
We will verify if IV injected ICG may colour breast tumors and axillary lymph nodes after neoadjuvant therapy (chemo- or hormonotherapy)

DETAILED DESCRIPTION:
In the operating room:

ICG 0.25 mg/kg will be given as an iv injection at least 20 minutes before the beginning of the operation.

Optionally, dynamic NIR imaging centered on the tumor bearing breast will be acquired during the 15 minutes after injection (in comparison with standards of known fluorescence intensity).

Optionally and in case of tumorectomy, peroperative "in vivo" imaging of the surgical dissection will be acquired. The tumour and/or the mammary piece (and the axillary piece) of dissection will be directly imaged "ex vivo" using the PDE camera (in comparison with standards of known fluorescence intensity).

In the Laboratory of Pathology:

The fresh mammary piece will be processed as usual, but the "gross-thick" sections will be imaged using the PDE and the fluorescent areas will be defined (and later analyzed in comparison with standards of known fluorescence intensity).

After fixation, the tumoral tissues as well as - if identified - non tumoral fluorescent foci will be thereafter processed "as usual".

All the slides obtained will be analyzed using the NIR fluorescent microscope for the presence or not of detectable ICG and the ICG-positive tissues or compartments (vascular spaces, interstitial spaces, normal and/or tumoral cells, macrophages…) will be determined.

If fluorescent foci are identified at the level of the axillary piece, they will be isolated and analyzed like the other lymph nodes. Using the NIR fluorescent microscope, these isolated macroscopically fluorescent structures will be analyzed (lymph node? Other?).

Additionally, metastatic lymph nodes will also be controlled for their microscopic fluorescence or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathological diagnosis of mammary cancer who have received neoadjuvant therapy and are candidate, either for tumorectomy, or for mastectomy with complete axillary node dissection,
* Informed consent form signed.

Exclusion Criteria:

* Diagnosis of mammary cancer established, either by tumorectomy, or by "gross" biopsy,
* Age less than18 years old.
* Inability to give informed consent.
* History of allergy or hypersensitivity against the investigational product (its active substance or ingredients), to iodine or to shellfish.
* Apparent hyperthyroidism, autonomous thyroid adenoma, unifocal, multifocal or disseminated autonomies of the thyroid gland.
* Documented coronary disease.
* Advanced renal impairment (creatinine > 1,5mg/dl).
* During the 2 weeks before the enrolment, concurrent medication which reduces or increases the extinction of ICG (i.e. anticonvulsants, haloperidol and Heparin).
* Pregnancy, breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
fluorescence intensity of tumoral lesions, scars and healthy tissues after IV injection of ICG in breast cancer patients after neoadjuvant therapy | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Veys, MD, Principal Investigator — Surgeon in Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Brussels Capital, Belgium